CLINICAL TRIAL: NCT00488033
Title: Screening For Asymptomatic Obstructive Coronary Artery Disease Among High-Risk Diabetic Patients Using CT Angiography, Following Core 64: A Randomized Control Study (The faCTor-64 Study)
Brief Title: Screening For Asymptomatic Obstructive Coronary Artery Disease Among High-Risk Diabetic Patients Using CT Angiography, Following Core 64
Acronym: faCTor-64
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Deseret Foundation (Other); Toshiba America Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 128-026
Record Dates: First submitted 2007-06-15; First posted 2007-06-19 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2014-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Diabetes; CT Angiography
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Standard of Care
- 2 (Other): CT Angiography
  Interventions: Procedure: CT Angiography

INTERVENTIONS:
Procedure: CT Angiography — If results indicate blockage, patients will receive interventional assessment (i.e., angiography) and treatment if indicated. All patients will receive aggressive treatment for type II diabetes (hemoglobin A1C) and lipids.
  Arms: 2

SUMMARY:
Patients with a known history of diabetes mellitus and no prior documented evidence of cardiovascular disease will be evaluated for inclusion in the study. Once qualified, patients will be enrolled and be randomized to either the Control Arm or to the Asymptomatic Screening Arm. Patients in the Control Arm will be followed by their primary care physicians with the recommendation that they follow standard guidelines for management of diabetic patients.

Patients in the Asymptomatic Screening Arm will undergo CT screening for either coronary calcium scoring or multi-slice CT angiography as well as be placed on one of two medical regimens. Patients will be followed by telephone at six-month intervals for a minimum of one year for both primary and secondary outcomes.

DETAILED DESCRIPTION:
Management of Patients Randomized to the Control Arm: Subjects randomized to the control arm will continue to be followed by their primary care physicians with the recommendation that they follow standard guidelines for management of diabetic patients.

Management of Patients Randomized to the Asymptomatic Screening Arm: Subjects randomized to the Asymptomatic Screening arm will undergo initial CT screening in the following fashion:

* Subjects with serum creatinine of < 2.0 mg/dl (men) or <1.8 mg/dL (women) will be screened using multi-slice CT angiography with contrast.
* Those with serum creatinine ≥ 2.0 mg/dl (men) or >1.8 mg/dL (women) will be screened without contrast to obtain a coronary calcium score. Further cardiac screening will be determined based on these results.

Subjects Receiving Multi-Slice CT Angiography (serum creatinine of < 2.0 mg/dl (men) or <1.8 mg/dL (women)): Subjects severe stenosis will proceed to coronary angiography and revascularization as needed. Subjects with moderate stenosis will be referred for adenosine stress cardiac MRI. If ischemia is detected, they will also be referred for coronary angiography. Subjects with either mild stenosis or normal coronary arteries will receive no further imaging studies.

Subjects Undergoing CT Evaluation for Coronary Calcium Scoring (serum creatinine ≥ 2.0 mg/dl (men) or >1.8 mg/dL (women): Subjects with coronary calcium scores >100 or >75th percentile will be referred for adenosine stress cardiac MRI. If ischemia is detected, they will be referred for coronary angiography. Subjects with coronary calcium scores = 0-10 or 11-100 and <75th percentile will receive no further imaging studies.

Medical Management (Only for those patients randomized to the Asymptomatic Screening Arm): In addition to the imaging studies and potential coronary revascularization procedures performed as described above, all subjects will be placed on one of two medical regimens:

* Standard Appropriate DM Care and
* Aggressive Risk Factor Reduction Care.

Standard Appropriate DM Care: Subjects assigned to this form of medical care will be managed by their primary physicians. This type of care will consist of targeting the goals proposed by Intermountain Healthcare for all patients with diabetes. These include the following three targets: HgA1C <7.0%, LDL cholesterol <100 mg/dL and Systolic BP<130 mm Hg. Subjects assigned to Standard Care will include all control subjects, as well as all screened subjects with either a normal CT angiogram or a coronary calcium score = 0-10.

Aggressive Risk Factor Reduction Care: Subjects assigned to this form of medical care, in addition to standard medical care provided by their primary physicians, will also be managed by their primary physicians, but will receive more aggressive risk factor reduction management according to a set of guidelines that will be given to the primary physicians. This aggressive management strategy, designed to address the increased medical risk among the asymptomatic diabetics with detected vascular disease, will consist of more aggressive glucose and lipid targets than is in the Standard Care protocols and specific medication algorithms designed to accomplish these more aggressive targets.

Follow-Up After enrollment into the protocol, all subjects will be followed for a minimum of one year. Follow-up will occur by telephone at six-month intervals. Outcomes will be ascertained by directly questioning the patient and by review of medical records. All primary outcomes will be adjudicated by an independent events committee.

Statistical Analysis Both an intention-to-treat analysis and a by protocol analysis will be performed. The intention-to-treat analysis will be the primary analysis and will be defined as all those randomized to scan versus all those randomized to control regardless of what actually happened. The by protocol analysis will be defined as all of those who actually got the protocol scan versus those who did not get the scan. Those who did not get the scan includes all those randomized to the control arm. If they went outside of the study and got a scan anyway, this will be considered to be for clinical indications and will still be in the non-protocol scan group. For those who were randomized to get the scan but never did, evaluation of their baseline characteristics will be made and if they did not differ from those who actually got the scan or from those who were randomized to control, then they will be included the didn't get scanned group.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Males ≥ 50 years; Females ≥55 years with: History of diabetes mellitus (prior documentation of fasting glucose ≥ 126 mg/dl or hemoglobin A1C > 6.5%), either type 1 or type 2, documented for at least 3 years and on medication for at least one year.
2. Age: Males ≥ 40 years; Females ≥45 years with: History of diabetes mellitus (prior documentation of fasting glucose ≥ 126 mg/dl or hemoglobin A1C > 6.5%), either type 1 or type 2, documented for at least 5 years and on medication for at least one year.
3. The patient or legally authorized representative must sign a written informed consent, prior to the procedure, using a form that is approved by the local Institutional Review Board.

Exclusion Criteria:

1. Known coronary artery disease (stenosis >70%, history of myocardial infarction, or angina)
2. Symptomatic cerebral vascular disease (history of TIA, CVA, or cerebrovascular [carotid or cerebral arteries] revascularization)
3. Symptomatic peripheral vascular disease (history of claudication, amputation, or peripheral [including renal arteries] arterial revascularization)
4. Treatment with any other investigational drug within the previous 30 days
5. Any therapy or condition that would pose a risk to the patient or make it difficult to comply with study requirements.
6. Pregnant and/or lactating women, and women of child bearing potential not using acceptable means of contraception. Women of childbearing potential must be using adequate measures of contraception (as determined by the Investigator) to avoid pregnancy and should be highly unlikely to conceive during the study period. Women of childbearing potential must have a negative pregnancy test at screen.
7. Any life threatening condition/significant co-morbidity such that primary screening is inappropriate.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2007-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Muhlestein, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Healthcare, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Muhlestein JB, Lappe DL, Lima JA, Rosen BD, May HT, Knight S, Bluemke DA, Towner SR, Le V, Bair TL, Vavere AL, Anderson JL. Effect of screening for coronary artery disease using CT angiography on mortality and cardiac events in high-risk patients with diabetes: the FACTOR-64 randomized clinical trial. JAMA. 2014 Dec 3;312(21):2234-43. doi: 10.1001/jama.2014.15825. PMID 25402757
- [Derived] Kwan AC, May HT, Cater G, Sibley CT, Rosen BD, Lima JA, Rodriguez K, Lappe DL, Muhlestein JB, Anderson JL, Bluemke DA. Coronary artery plaque volume and obesity in patients with diabetes: the factor-64 study. Radiology. 2014 Sep;272(3):690-9. doi: 10.1148/radiol.14140611. Epub 2014 Apr 22. PMID 24754493

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Managed by primary care physicians with recommendation to follow the guidelines for standard appropriate diabetes care.
- Coronary Computed Tomographic Angiography: Received medical management recommendations based on the results of their CT scans.
Period: Overall Study
Arm/Group | Standard of Care | Coronary Computed Tomographic Angiography
Started | 448 | 452
Completed | 447 | 452
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Coronary Computed Tomographic Angiography | Total
Number analyzed (Participants) | 447 | 452 | 899
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (8.35) | 61.5 (7.94) | 61.5 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 218 | 430
  Male | 235 | 234 | 469
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 427 | 434 | 861
  Hispanic | 13 | 10 | 23
  African American | 1 | 2 | 3
  Asian | 3 | 2 | 5
  American Indian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.4 (7.05) | 32.9 (6.76) | 33.1 (6.90)
Smoking History or Current [Count of Participants; unit: Participants] | 68 | 75 | 143
Diabetes Mellitus [Mean (Standard Deviation); unit: years] | 13.5 (10.72) | 12.3 (9.23) | 12.9 (10.01)
Diabetes Mellitus Type [Count of Participants; unit: Participants]
  Type I | 52 | 56 | 108
  Type II | 395 | 396 | 791
Diabetes Mellitus Medications [Count of Participants; unit: Participants]
  Non-Insulin Agent Only | 255 | 258 | 513
  Insulin Only | 95 | 84 | 179
  Both Non-Insulin Agent and Insulin | 97 | 110 | 207
Hemoglobin A1C [Mean (Standard Deviation); unit: percentage] | 7.5 (1.41) | 7.4 (1.40) | 7.5 (1.41)
Hemoglobin A1C Category [Count of Participants; unit: Participants] — Population: Hemoglobin A1C information was unavailable for 40 participants.
  Participants
    number analyzed (Participants) | 431 | 428 | 859
    ≤ 6.5 | 101 | 120 | 221
    6.5-8.0 | 225 | 210 | 435
    >8.0 | 105 | 98 | 203
Family History of Diabetes Mellitus [Count of Participants; unit: Participants] | 59 | 44 | 103
Family History of Cardiovascular Disease [Count of Participants; unit: Participants] | 88 | 69 | 157
Hypertension [Count of Participants; unit: Participants] | 308 | 287 | 595
Hyperlipidemia [Count of Participants; unit: Participants] | 282 | 285 | 567
Hypothyroidism/Hyperthyroidism [Count of Participants; unit: Participants] | 104 | 104 | 208
Depression [Count of Participants; unit: Participants] | 58 | 59 | 117
Gastroesophageal Reflux DIsease [Count of Participants; unit: Participants] | 98 | 92 | 190
Sleep Apnea [Count of Participants; unit: Participants] | 115 | 121 | 236
Asthma [Count of Participants; unit: Participants] | 48 | 45 | 93
Arthritis [Count of Participants; unit: Participants] | 11 | 8 | 19
Renal DIsease [Count of Participants; unit: Participants] | 32 | 33 | 65
Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 130.5 (11.49) | 129.1 (12.45) | 129.8 (12.00)
  Diastolic | 74.1 (7.71) | 74.2 (8.41) | 74.1 (8.06)
Statin Use [Count of Participants; unit: Participants] | 322 | 346 | 668
Fasting Lipid Panel [Mean (Standard Deviation); unit: mg/dL]
  LDL cholesterol | 87.7 (32.92) | 86.3 (29.12) | 87.0 (31.07)
  HDL cholesterol | 45.3 (13.41) | 45.4 (14.04) | 45.3 (13.72)
Fasting Triglycerides [Median (Inter-Quartile Range); unit: mg/dL] | 132 [92 to 198] | 144 [99 to 201] | 139 [96 to 200]
LDL Cholesterol Categories [Count of Participants; unit: Participants] — Population: LDL category was unavailable for 82 participants.
  Participants
    number analyzed (Participants) | 409 | 408 | 817
    ≤70 | 124 | 123 | 247
    70-100 | 179 | 169 | 348
    >100 | 106 | 116 | 222
Creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 0.92 [0.80 to 1.10] | 0.91 [0.79 to 1.10] | 0.91 [0.80 to 1.10]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Combination of All Cause Death, Non-fatal Myocardial Infarction (MI), and Hospitalization for Unstable Angina
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Coronary Computed Tomographic Angiography
Number analyzed (Participants) | 447 | 452
Participants | 34 | 28

2. Secondary Outcome: Number of Participants Suffering Cardiovascular (CV) Death
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Coronary Computed Tomographic Angiography
Number analyzed (Participants) | 447 | 452
Participants | 8 | 7

3. Secondary Outcome: Number of Participants With Combination of Coronary Death, Non-fatal MI, and Unstable Angina With Hospitalization
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Coronary Computed Tomographic Angiography
Number analyzed (Participants) | 447 | 452
Participants | 23 | 21

4. Secondary Outcome: Number of Participants With Hospitalization for Heart Failure
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Coronary Computed Tomographic Angiography
Number analyzed (Participants) | 447 | 452
Participants | 10 | 3

5. Secondary Outcome: Number of Participants With Stroke or Carotid Revascularization Procedure
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Coronary Computed Tomographic Angiography
Number analyzed (Participants) | 447 | 452
Participants | 9 | 8

6. Secondary Outcome: Number of Participants With Limb Amputation or Peripheral Vascular Revascularization Procedure
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Coronary Computed Tomographic Angiography
Number analyzed (Participants) | 447 | 452
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: 2-7 years (mean 4 years)
Arm/Group | Standard of Care | Coronary Computed Tomographic Angiography
All-Cause Mortality (participants affected / at risk) | 19/447 | 16/452
Serious Adverse Events (participants affected / at risk) | 28/447 | 29/452
Other Adverse Events (participants affected / at risk) | 0/447 | 0/452
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=447) | Coronary Computed Tomographic Angiography (N=452)
Non-Fatal MI (Cardiac disorders) | 8 (8) | 7 (7)
Hospitalization for Unstable Angina (Cardiac disorders) | 9 (9) | 9 (9)
Hospitalization for Heart Failure (Cardiac disorders) | 10 (10) | 3 (3)
Stroke or Carotid Revascularization Procedure (Vascular disorders) | 9 (9) | 8 (8)
Limb Amputation or Peripheral Vascular Revascularization Procedure (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes